CLINICAL TRIAL: NCT00852800
Title: Effect of Intravenous Albumin (Standard vs Dose Reduced Regimen) On Renal Impairment and Mortality in Patients With Cirrhosis and Spontaneous Bacterial Peritonitis: A Double Blind Randomized Clinical Trial
Brief Title: Low-dose Albumin Solution in SBP: a Randomized Double-blind Pilot Study
Acronym: ALTERNATE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Mário Reis Álvares-da-Silva, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-352
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Renal Impairment; All Cause Mortality
Keywords: spontaneous bacterial peritonitis; albumin; renal impairment; mortality
MeSH Terms: conditions — Renal Insufficiency | interventions — Albumins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard regimen (Active Comparator): Albumin in standard regimen (1.5 g/Kg IV on day 1 and 1 g/kg IV on day 3)with saline solution to complete total volume of 1000 ml on day 1 and 500 ml on day 3
  Interventions: Drug: Albumin
- Dose reduced regimen (Experimental): Albumin in dose reduced regimen (1 g/kg IV on day 1 and 0.5 g/kg IV on day 3) with saline solution to complete total volume of 1000 ml on day 1 and 500 ml on day 3
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Albumin — 1.5 g/kg IV on day 1 and 1 g/kg IV on day 3 with saline solution to complete total volume of 1000 ml on day 1 and 500 ml on day 3. Infusion in 4 hours.
  Other Names: Albumin at standard dose diluted with saline solution
  Arms: Standard regimen
Drug: Albumin — 1 g/kg IV on day 1 and 0.5 g/kg IV on day 3 with saline solution to complete total volume of 1000 ml on day 1 and 500 ml on day 3. Infusion in 4 hours.
  Other Names: Albumin at dose reduced diluted with saline solution
  Arms: Dose reduced regimen

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a common and severe complication of cirrhosis. The most serious complication of SBP is the hepatorenal syndrome (HRS), which occurs in up to 30 percent of patients, with high mortality. Intravenous albumin (1.5 g/kg at diagnosis and 1 g/kg 48 hours later - standard regimen) helps to prevent HRS and improves survival. No information exists on the efficacy of lower doses of albumin. This study was designed to allow direct comparison among different doses of intravenous albumin in patients with SBP - standard (SR) vs dose reduced regimen (DRR) - in order to prevent renal failure and mortality.

DETAILED DESCRIPTION:
Patients with cirrhosis who had spontaneous bacterial peritonitis (SBP) and who are admitted from March 2006 to a single university hospital were evaluated for inclusion in the study. The study was approved by the investigational review boar, and patients gave written informed consent to participate. Inclusion criteria were a cytological diagnosis of SBP, in the absence of findings suggestive of secondary peritonitis; age between 18 and 80 years; no antibiotic treatment within one week before the diagnosis of spontaneous bacterial peritonitis (except for prophylactic treatment with norfloxacin or trimethoprim/sulfamethoxazole); the absence of other infections, shock, gastrointestinal bleeding, grade 3 or 4 hepatic encephalopathy, cardiac failure, and any disease (e.g., advanced neoplasia) that could affect the short term prognosis; a serum creatinine level of no more than 3 mg per deciliter 265 µmol per liter); and the absence of potential causes of dehydration (such as diarrhea or an intense response to diuretic treatment) within one week before the diagnosis of peritonitis.

Patients were randomly assigned to one of two groups: standard regimen (SR) vs dose reduced regimen (DRR). Randomization was performed independently with the use of sealed envelopes containing the treatment assignments, which were based on random numbers generated by computer. All the investigators were unaware of the treatment assignments.

Physical examination and routine laboratory tests (blood-cell counts and liver and renal tests) and measurement of plasma rennin activity were performed on day 1 of therapy in all patients. Laboratory measurements were repeated every three days until discharge. Rennin activity was repeated on day 7. Intravenous cefotaxime was given daily in doses that varied accordingly to creatinine. Albumin was given at a dose of 1.5 or 1 g per kilogram of body weight on day 1, followed by 1 or 0.5 g per kilogram on day 3 (SR vs DRR). Albumin was diluted in saline solution until total volume of 1000 ml on day 1 and 500 ml on day 3. Albumin was prepared in a bottle with same color, volume and aspect in both groups. Diuretic treatment was not give until day 5 of treatment and therapeutic paracentesis > 3 liters was not allowed until the infection had resolved. Response to cefotaxime was considered when the polymorphonuclear-cell count in ascitic fluid reduced by at least 50%. Antibiotic treatment was modified when no response to cefotaxim occurred according to the in vitro susceptibility of the isolated organism or was modified empirically in patients with negative blood and ascitic-fluid cultures. Prophylactic norfloxacin or trimethoprim/sulfamethoxazole therapy was initiated after the resolution of infection and was maintained throughout the follow-up period. Renal failure at the time of enrollment was diagnosed when the serum creatinine level was more than 1.5 mg per deciliter. Renal impairment was defined as a nonreversible deterioration of renal function during hospitalization. In patients without renal failure at enrollment, renal impairment was diagnosed when serum creatinine level increased by more than 50 percent of the pretreatment value, to level higher than 1.5 mg per deciliter. In patients with preexisting renal failure, an increase in serum creatinine level by more than 50 percent from base line was required for a diagnosis of renal impairment. After the resolution of infection, patients with tense ascites were treated with total paracentesis and the administration of albumin, regardless of treatment assignment, followed by sodium restriction and diuretic therapy, and those with moderate ascites were treated only with sodium restriction and diuretics. After discharge from the hospital, patients were followed until 90 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* cytological diagnosis of spontaneous bacterial peritonitis
* age between 18 and 80 years
* written informed consent

Exclusion Criteria:

* findings suggestive of secondary peritonitis
* antibiotic treatment within one week before the diagnosis of spontaneous bacterial peritonitis (except for prophylactic treatment with norfloxacin or trimethoprim/sulfamethoxazole)
* other infections, shock, gastrointestinal bleeding, grade 3 or 4 hepatic encephalopathy, cardiac failure, and any disease (e.g., advanced neoplasia) that could affect the short term prognosis
* creatinine level of more than 3 mg per deciliter
* potential causes of dehydration (such as diarrhea or an intense response to diuretic treatment) within one week before the diagnosis of peritonitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-03; Primary Completion 2009-08 (Actual); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
renal impairment | within first 90 days
all cause mortality | within first 90 days

SECONDARY OUTCOMES:
Plasmatic renin activity | day 0 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Mário R Álvares-da-Silva, Principal Investigator — Hospital de Clínicas de Porto Alegre; Alexandre Araujo, Study Chair — Hospital de Clínicas de Porto Alegre; Gabriela Rossi, Study Chair — Hospital de Clínicas de Porto Alegre; Antônio B Lopes, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil